CLINICAL TRIAL: NCT07250945
Title: Study of the Effectiveness of the ADVATx Laser in the Treatment of Port-wine Stains
Brief Title: AdvaTx Laser Treatment for Vascular Birthmarks
Acronym: ADVA-PWS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Kemény Lajos, Professor, MD, DSc, MHAS, Szeged University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD-ADVA-01; CIV-HU-25-08-053915 (Other: National Centre for Public Health and Pharmacy, Budapest)
Record Dates: First submitted 2025-09-23; First posted 2025-11-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Port-wine Stains (PWS); Vascular Birthmark
Keywords: ADVATx laser; Port-wine stain; Vascular Birthmark
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AdvaTx laser treated (Other): AdvaTx laser treated patients
  Interventions: Device: ADVATx laser treatment

INTERVENTIONS:
Device: ADVATx laser treatment — Patients in the study will receive ADVATx laser treatment (1 treatment per month for 4 months) The treatment takes approximately 10-30 minutes per session. The treatment lasts for a total of 5 months for one patient. At each treatment session photographic documentation will be performed. PRO will be assessed by a questionnaire. At the end of the study, the patient rates the treatment and improvement on a Patient Satisfaction Scale.

SUMMARY:
The primary objective of the present study is to get experiences with the use of CE-marked ADVATx laser treatment for port-wine stains.

Secondary objectives: To investigate the clinical efficacy of ADVATx laser treatment for port-wine stains.

To investigate the potential side effects (erythema, hyperpigmentation, oedema, pain, swelling, skin burning, blisters) of the treatment.

Patients in the study will receive ADVATx laser treatment (1 treatment per month for 4 months) The treatment takes approximately 10-30 minutes per session. The treatment lasts for a total of 5 months for one patient. At each treatment session photographic documentation will be performed. PRO will be assessed by a questionnaire. At the end of the study, the patient rates the treatment and improvement on a Patient Satisfaction Scale.

DETAILED DESCRIPTION:
Prospective testing and evaluation of a ADVATx, a CE marked device within its intended use, carried out in one centre.

The ADVATx™ laser system, a solid-state laser with wavelengths of 589 nm and 1319 nm. It offers a solution for an exceptionally wide range of indications. It can treat more than 15 indications related to vascular lesions and other dermatological problems with excellent results and high patient safety. It is extremely economical to operate.

Only medical personnel qualified to use medical lasers are authorised to use them.

EUDAMED registration

Advalight card with SRN number:

https://ec.europa.eu/tools/eudamed/#/screen/search-eo/8de1b38d-a0dc-4315-b068-3416928deabe Actor ID/SRN: DK-MF-000010334 Classification of ADVATx: Class IIb medical device

ELIGIBILITY:
Inclusion Criteria:

1. The patient understands the information provided, gives informed consent to participate in the study and is deemed by the investigator to be able to participate,
2. a signed consent form,
3. parental consent is required for patients under 18 years of age,
4. the lesions to be treated are at least 15 cm2,
5. the study is open to Fitzpatrick skin types I-IV.

Exclusion Criteria:

1. Lack of parental consent for patients under 18 years of age,
2. symptoms localised to the central part of the face (cheeks, nose),
3. people with Fitzpatrick skin type V-VI,
4. pregnancy,

4. epilepsy, 5. fever, infectious diseases, 6. the patient is within one month or currently enrolled in another clinical trial.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in lesion presentation measured by Investigator Global Assessment (IGA) | 5 months
  The IGA is a five-point scale from 0 (no change) to 4 (complete or nearly complete clearance). Three blinded dermatologists will review standardized clinical photographs to evaluate each treated area. Results will be reported as the average IGA score for each treatment method.

SECONDARY OUTCOMES:
Patient satisfaction score | 5 months
  Patients will rate their satisfaction with the treated area using a 0-6 scale, where 0 indicates no satisfaction and 6 indicates very satisfied.
Pain score during laser treatment measured by Visual Analog Score (VAS) | 5 months
  Participants will assess their pain during each treatment using a Visual Analog Scale (VAS), which ranges from 0 (no pain) to 10 (the worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Albert Szent-Györgyi Clinical Centre, Department of Dermatology and Allergology, Szeged, Csongrád-Csanád Vármegye, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clinicians Rely on ADVATx for Acne Scars and Unwanted Vascularity By Kevin A. Wilson, Contributing Editor THE Aesthetic Guide May/June 2018 www.aestheticchannel.com
- [Background] Next-Generation ADVATx Platform Transcends Pulsed Dye Lasers By Kevin A. Wilson, Contributing Editor The Aesthetic Guide March/April 2018 www.aestheticchannel.com